CLINICAL TRIAL: NCT00490633
Title: Reducing the Transmission of Influenza by Face Masks
Brief Title: Intervention Study of Face Mask and Hand Sanitizer to Reduce Influenza Transmission
Acronym: M-FLU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Arnold S. Monto, University of Michigan
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: HUM00008566
Record Dates: First submitted 2007-06-21; First posted 2007-06-25 (Estimated); Last update posted 2011-08-19 (Estimated); Status verified 2007-06

CONDITIONS: Influenza
Keywords: Influenza; Non Pharmaceutical Intervention; Face Mask; Hand Hygiene
MeSH Terms: conditions — Influenza, Human | interventions — Ethanol; Hand Sanitizers

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Facemask and hand hygiene (Experimental): Facemask and hand hygiene provided for participants.
  Interventions: Behavioral: Ear Loop Procedure Mask; Behavioral: 62% Ethyl Alcohol Hand Sanitizer
- Facemask only (Experimental): Facemask only provided for participants.
  Interventions: Behavioral: Ear Loop Procedure Mask
- Control (No Intervention): Control, no intervention.

INTERVENTIONS:
Behavioral: Ear Loop Procedure Mask — Facemasks were requested to be worn while participants were in the residence hall for year one, and while they were in residence halls for a minimum of six hours per day in year two.
  Other Names: TECNOL™ procedure masks, Kimberly-Clark, Roswell GA
  Arms: Facemask and hand hygiene; Facemask only
Behavioral: 62% Ethyl Alcohol Hand Sanitizer — Hand sanitizer was provided to participants in the facemask and hand hygiene arm for year one and year two of the study.
  Other Names: Purell, 62% ethyl alcohol in a gel base
  Arms: Facemask and hand hygiene

SUMMARY:
Pharmaceutical interventions, particularly vaccination, have been the principal public health method of preventing and controlling seasonal influenza. Other less invasive non-pharmaceutical interventions include the use of face masks and hand hygiene. In Asia, masks are used extensively, especially in Japan, but with only circumstantial evidence of efficacy. Although there are numerous studies that support hand hygiene as an effective measure for decreasing transmission of enteric infections, there are fewer data assessing the effect of hand hygiene on respiratory illnesses. Therefore it is proposed that a study be conducted on the use of face masks with and without the use of hand hygiene in comparison to no intervention in residence housing units of the University of Michigan. The interventions will be carried out during a period of influenza transmission that is defined by surveillance conducted at the University Health Service. Data will be collected on use of the interventions and the occurrence of influenza and other illnesses. When illness occurs meeting a case definition, specimens for viral isolation will be collected in all intervention settings. Face masks could theoretically lead to a large reduction in transmission frequency of influenza, especially if most transmission occurs by the airborne (large or small droplet) route. Even a modest reduction could have a major effect during an influenza pandemic.

DETAILED DESCRIPTION:
Objective:

The overall objective of this study is to investigate the feasibility and effectiveness of various non-pharmaceutical interventions on the occurrence of influenza in residence units of the University of Michigan.

Specific Aims:

The three specific aims of this study are to: (1) determine the feasibility of using face masks and hand hygiene education among students living in residence hall units at the University of Michigan, (2) estimate the reduction of influenza infection and illness during laboratory documented influenza outbreaks in individuals and groups using one or more interventions compared to those not using such interventions, and (3) track occurrence of influenza cases in the participating residence units of the University.

Background:

Community based intervention studies that target prevention of droplet transmission, via face masks in addition to hand-to-hand transmission along with alcohol-based antiseptic use, are needed along with culture confirmed respiratory illness data.

Methodology:

The proposed study is a randomized intervention designed to examine the effectiveness of face masks alone and layered face masks and hand hygiene interventions for reducing transmission of influenza among students residing in University of Michigan residence halls during laboratory defined influenza seasons. Randomization will be by geographically separate housing unit. In the first year, residence halls will be assigned to each of the interventions and to the observed comparison to bring the total number of participants to 750 in each of the interventions and the comparison (total number: 2250). For year two, randomization was performed at the residence house level to increase clustering units and also aimed for 750 students in each intervention. Students living in each of the residence halls will be asked if they wish to participate in the study. Those giving informed consent will be asked to complete a survey each week to ascertain illness occurrences. When influenza illness is documented to be occurring in the University setting, the interventions will be implemented. During that period, the survey will be expanded to include questions on intervention use, as appropriate for the particular housing unit. Also during this period, those with illnesses meeting a case definition will be asked to provide specimens for virus identification. This collection will not be limited to those agreeing to the use of the interventions, since informed consent will be obtained for all specimen collections.

Intervention Methods:

Randomization will be clustered by residence hall since it is likely that incidence of influenza infection will be correlated among subjects within residence halls. In year 2, clustering was done by residence house to increase the clustering units. The intervention residence halls will receive one of the following two interventions: (i) masks alone or (ii) masks plus alcohol-based hand sanitizers (62% ethyl alcohol) and hygiene education. The remaining halls will serve as comparison units. The control dorms will be similar to the intervention dorms on basic demographic distributions, such as age range and geographical proximity. Residence halls that are randomized to the control arm will not receive any masks, hygiene education materials, or alcohol-based hand sanitizer.

Within each of the randomized residence halls assigned to receive an intervention, our goal is to assess the use of face masks and hand sanitizer. The intervention will be put into effect only when two or more virus positive illnesses are detected in a single week. Rapid tests will be available to help in identifying cases if laboratory confirmation may be delayed. The use of face masks will continue until the outbreak is recognized by virology to be coming to a close or after the passage of 6 weeks, whichever occurs first. It is felt that there needs to be a guaranteed duration in order to assure compliance with face mask use.

Face Mask:

Residence halls receiving interventions (i) and (ii) will receive face masks and will be asked to comply with their use at least while in the residence hall when it is known that influenza virus is transmitting on campus. A week's supply of face masks and plastic bags for disposal will be bundled along with instructions for use. They will be requested to wear the masks when out of the halls, but this may be more difficult to implement. As indicated below, we will ask what proportion of time the masks are worn. The choice of the specific face masks will be carried out in conjunction with the CDC project officers. The face mask intervention would require a once a day change during use to ensure proper protection and a hygienic barrier. It is clear from the recent Institute of Medicine report that little is known about long term use or reuse of face masks, so variations in the number of times in which a face mask is changed is a variable that could be assessed in this study.

The use of face masks will continue for 6 weeks. Instructions will be given as to the correct and incorrect way to utilize surgical masks. As part of the evaluation of level of use, staff observers in each facility will estimate what proportion of individuals actually use them properly. This will take place in common rooms, hallways, and residence hall dining facilities to supplement the self reports that will be collected by e-mail from all participants.

Hand Hygiene Education and Antiseptic Product Use:

All students in residence halls receiving intervention (ii) will be provided with a comprehensive hand hygiene education component in addition to mask use. The educational component will include posters and pamphlets that provide background information on transmission of influenza, an explanation of the effectiveness of hand hygiene for reducing transmission, and guidelines for proper hand hygiene, including the need for hand hygiene at critical locations throughout the residence halls. The hand washing campaign will consist of posters on bulletin boards and weekly email hand hygiene reminder messages to participants in the intervention residence halls. The educational component of the study will include a video for both the control arm and the intervention arms. The control video will address information on influenza and an overview of the study. The intervention video will address both information on influenza and an overview of the study, in addition to hand hygiene education and the use of hand sanitizer and the use of face masks. Both videos are available on the website (www.mflu.org) and on Survey Monkey linked to the consent form.

The intervention dorms will be given a portable alcohol-based hand sanitizer and a large stationary pump alcohol-based hand sanitizer to use throughout the study period in addition to basic hand hygiene education materials and messages. In order to quantify the effect of the alcohol-based hand sanitizer use on influenza virus transmission, regular self reports of hand-sanitizer use will be collected and the products provided will be monitored for use (by weighing) and re-supplied as needed on a weekly basis during the influenza season. Control participants will also be required to provide information on type and name of product used and daily frequency of use, should they be using any.

Control Residence Halls:

Students residing in the control housing units will be asked to participate in the disease surveillance aspect of the study. They will be contacted by e-mail, be asked to consent to participate in a wellness study in which they will report on respiratory and enteric illness symptoms on a weekly basis. The students will be compensated for this participation but not at the level of those who are in the intervention arms.

Hand Hygiene, Face Mask and Illness Surveillance:

Participants in both the intervention and control housing units will be asked to report information on a weekly basis concerning use of the interventions (where appropriate) and the occurrence of respiratory and enteric illness symptoms. Questions on the health attitudes and knowledge will be collected at the start and end of the study season. This survey will be modified for residence hall participants so that frequency of use of face masks can be similarly determined, including attitudes about wearing them.

Both intervention compliance and outcome measures will be collected via electronic survey. This will include mask use, alcohol-based hand sanitizer use, and details regarding respiratory symptoms and enteric symptoms. During the first year, the survey instruments will be assessed for reliability for use among our target student populations in residence halls and may be modified in the second year. Honoraria will be calculated based on the weeks the report is completed, and paid at the end of the season.

Collection of Specimens for Virus Identification:

All residents in the intervention and comparison residences will receive small magnetic cards, modified after those currently used in the vaccine study, describing the case definition. An individual will be asked to have a specimen collected for virus identification whenever an illness that meets the case definition occurs. Information on symptoms, duration of illnesses and other relevant characteristics will be obtained.

Laboratory Methods for Virus Identification:

All specimens for virus identification will be collected by throat swab and placed in veal infusion broth transport medium. This transport medium has been found to protect viruses for days during shipment from remote sites and to be suitable for PCR tests as well.

Positives are passed to additional tubes of cell culture. Initial typing is carried out by fluorescent antibody techniques. Subtyping of type A viruses are carried out by hemagglutination-inhibition. For specimens collected in the influenza vaccine efficacy study, specimens are also processed by real time PCR. By collecting data on vaccination use among participants, we will be able to control for vaccine use in our study analyses. Given the low rate of vaccination uptake among college age individuals, we do not expect vaccine use to be a significant confounder in our study design.

Statistical Design:

To estimate the reduction of influenza infection and illness during laboratory documented influenza outbreaks in individuals and groups using one or more interventions compared to those not using such interventions. The effect of the intervention will be tested through the use of generalized estimating equations (GEE) as applied to statistical regression models for clustered data. The main outcome for this aim will be the rate of influenza cases and rates of secondary influenza transmission comparing the intervention and control dormitories. Additional outcomes will include other non-influenza respiratory illnesses and enteric illness symptoms. Predictor variables will include the main effects of the intervention and control for potential confounders depending upon balance of the known confounders across intervention and control residence halls.

ELIGIBILITY:
Inclusion Criteria:

* Residence in selected University of Michigan Residence Halls

Exclusion Criteria:

* Non-residence in selected Residence Halls
* Unwillingness to utilize face mask and hand sanitizer and complete online surveys
* Already study employee

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1420 (Actual)
Dates: Start 2006-10; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Number of laboratory confirmed cases of Influenza | 8 weeks, including the 6 weeks of intervention and two weeks post-intervention

SECONDARY OUTCOMES:
Number of cases of Influenza Like Illness | 6 weeks of intervention

CONTACTS AND LOCATIONS:
Overall Officials: Arnold S Monto, MD, Principal Investigator — University of Michigan; Allison E Aiello, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

REFERENCES:
- [Result] Aiello AE, Murray GF, Perez V, Coulborn RM, Davis BM, Uddin M, Shay DK, Waterman SH, Monto AS. Mask use, hand hygiene, and seasonal influenza-like illness among young adults: a randomized intervention trial. J Infect Dis. 2010 Feb 15;201(4):491-8. doi: 10.1086/650396. PMID 20088690
- [Derived] Jefferson T, Dooley L, Ferroni E, Al-Ansary LA, van Driel ML, Bawazeer GA, Jones MA, Hoffmann TC, Clark J, Beller EM, Glasziou PP, Conly JM. Physical interventions to interrupt or reduce the spread of respiratory viruses. Cochrane Database Syst Rev. 2023 Jan 30;1(1):CD006207. doi: 10.1002/14651858.CD006207.pub6. PMID 36715243
- [Derived] Jefferson T, Del Mar CB, Dooley L, Ferroni E, Al-Ansary LA, Bawazeer GA, van Driel ML, Jones MA, Thorning S, Beller EM, Clark J, Hoffmann TC, Glasziou PP, Conly JM. Physical interventions to interrupt or reduce the spread of respiratory viruses. Cochrane Database Syst Rev. 2020 Nov 20;11(11):CD006207. doi: 10.1002/14651858.CD006207.pub5. PMID 33215698
- [Derived] Aiello AE, Perez V, Coulborn RM, Davis BM, Uddin M, Monto AS. Facemasks, hand hygiene, and influenza among young adults: a randomized intervention trial. PLoS One. 2012;7(1):e29744. doi: 10.1371/journal.pone.0029744. Epub 2012 Jan 25. PMID 22295066
- [Derived] Perez V, Uddin M, Galea S, Monto AS, Aiello AE. Stress, adherence to preventive measures for reducing influenza transmission and influenza-like illness. J Epidemiol Community Health. 2012 Jul;66(7):605-10. doi: 10.1136/jech.2010.117002. Epub 2011 Jan 10. PMID 21224242